CLINICAL TRIAL: NCT01001949
Title: In Vivo Evaluation of the Physiological Effects of Arabinoxylan-oligosaccharides (AXOS) in Healthy Subjects: a Randomized, Placebo-controlled, Double-blind, Cross-over Study
Brief Title: In Vivo Evaluation of the Physiological Effects of Arabinoxylan-oligosaccharides (AXOS) in Healthy Subjects (Juniors)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fugeia NV (Industry)
Responsible Party: Kristin Verbeke, Ph.D., Katholieke Universiteit Leuven
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ML5282 junior
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Gastrointestinal Health; Healthy Subjects
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wheat Bran Extract (Experimental)
  Interventions: Dietary Supplement: Wheat Bran Extract
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Wheat Bran Extract — soft drink comprising WBE and natural flavor and coloring agent, ingestion after breakfast and after dinner
  Arms: Wheat Bran Extract
Dietary Supplement: placebo — soft drink with natural flavor and coloring agent, without WBE, ingestion after breakfast and dinner
  Arms: placebo

SUMMARY:
The investigational product used in this study is a soft drink containing an arabinoxylan-oligosaccharide (AXOS) preparation extracted from wheat bran (hereafter called Wheat Bran Extract, WBE).

The objective of this study is to analyze the effect of the intake of WBE on various parameters of gastrointestinal health in children (8-12 yrs). Additionally, safety was analyzed using treatment emergent Adverse Events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* regular eating habits
* consent to take in the study product according to the study protocol
* consent of parents for follow-up of the protocol
* subject is willing to maintain his/her habitual food and beverage intake throughout the study period (with the exception of omission of prebiotic and probiotic food products as indicated in the study protocol)

Exclusion Criteria:

* low-calorie diet or other extreme dietary habits in the 6 weeks before the start of the clinical trial
* recent use of antibiotics
* abdominal surgery in the past
* use of medication or dietary supplements known to influence gastrointestinal tract within two weeks of start of clinical trial. Examples of such medication/dietary supplements are antispasmodics, anti-diarrhea medication and/or probiotic medication
* serious illness within 3 months of start of clinical trial
* chronic gastrointestinal conditions such as inflammatory bowel disease (IBD), irritable bowel syndrome (IBS), chronic constipation, history of frequent diarrhea, clinically important lactose intolerance
* complete anesthetics within 3 month of the start of the clinical trial
* allergy for wheat products
* celiac disease
* Subject has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the subject at undue risk

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Bifidobacteria content in feces | day 19 or 20 of each intervention period
butyric acid content in feces | day 19 or 20 of each intervention period
stool frequency | third week of each intervention period

SECONDARY OUTCOMES:
adverse events | whole study period

CONTACTS AND LOCATIONS:
Overall Officials: Willem Broekaert, Ph.D., Study Director — Fugeia NV
Locations (1):
- Department of Gastrointestinal Research, Laboratory Digestion and Absorption, Leuven, Belgium

REFERENCES:
- [Derived] Francois IE, Lescroart O, Veraverbeke WS, Marzorati M, Possemiers S, Hamer H, Windey K, Welling GW, Delcour JA, Courtin CM, Verbeke K, Broekaert WF. Effects of wheat bran extract containing arabinoxylan oligosaccharides on gastrointestinal parameters in healthy preadolescent children. J Pediatr Gastroenterol Nutr. 2014 May;58(5):647-53. doi: 10.1097/MPG.0000000000000285. PMID 24368315